CLINICAL TRIAL: NCT04888715
Title: An Open Label, 2-part, One-sequence, 3-period Study to Evaluate Drug-drug Interactions Between "DWN12088" and "Pirfenidone" or "Nintedanib" in Healthy Volunteers
Brief Title: To Evaluate Drug-drug Interactions Between DWN12088 and Pirfenidone or Nintedanib in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DW_DWN12088103
Record Dates: First submitted 2021-04-28; First posted 2021-05-17 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — pirfenidone; nintedanib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DWN12088 and Pirfenidone (Experimental): T1 - Pirfenidone A mg, Tablet, oral, once daily, T2 - 1) DWN12088 X mg, Tablet, oral, once daily, 2) DWN12088 X mg, Tablet, oral, twice daily, T3 - DWN12088 X mg, Tablet, oral, once daily+ Pirfenidone A mg, Tablet, oral, once daily
  Interventions: Drug: DWN12088; Drug: Pirfenidone
- DWN12088 and Nintedanib (Experimental): T1 - Nintedanib B mg, Tablet, oral, once daily, T2 - DWN12088 X mg, Tablet, oral, twice daily, T3 - DWN12088 X mg, Tablet, oral, once daily+ Nintedanib B mg, Tablet, oral, once daily
  Interventions: Drug: DWN12088; Drug: Nintedanib

INTERVENTIONS:
Drug: DWN12088 — Prolyl-tRNA synthetase (PRS) inhibitor
Drug: Pirfenidone — Pirfenidone
  Arms: DWN12088 and Pirfenidone
Drug: Nintedanib — Nintedanib
  Arms: DWN12088 and Nintedanib

SUMMARY:
An open label, 2-part, one-sequence, 3-period study to evaluate drug-drug interactions between DWN12088 and Pirfenidone or Nintedanib in healthy volunteers

DETAILED DESCRIPTION:
This clinical trial is an open label, 2-part, one-sequence, 3-period study to evaluate drug-drug interactions between DWN12088 and Pirfenidone or Nintedanib in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged ≥ 19 and ≤ 55 years at screening
* Subjects who voluntarily decided to participate in the study and provided written consent to after receiving a detailed explanation on this study and fully understanding the information

Exclusion Criteria:

* Subjects who received another investigational agent in another study (including bioequivalence study) within 180 days prior to the first dose of the IP (The end of prior study participation will be the date of the last dose, and the days will be counted from the next day [1 day].)
* Female subjects who are pregnant or lactating

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2021-07-23 (Actual); Primary Completion 2021-08-02 (Actual); Study Completion 2021-08-18 (Actual)

PRIMARY OUTCOMES:
Cmax of Pirfenidone and DWN12088 | 0hour (pre-dose), 1hour, 2hour, 3hour, 4hour, 6hour, 8hour, 10hour, 12hour
  Cmax of Pirfenidone and DWN12088
AUC of Pirfenidone and DWN12088 | 0hour (pre-dose), 1hour, 2hour, 3hour, 4hour, 6hour, 8hour, 10hour, 12hour
  AUC of Pirfenidone and DWN12088
Cmax of Nintedanib and DWN12088 | 0hour (pre-dose), 1hour, 2hour, 3hour, 4hour, 6hour, 8hour, 10hour, 12hour
  Cmax of Nintedanib and DWN12088
AUC of Nintedanib and DWN12088 | 0hour (pre-dose), 1hour, 2hour, 3hour, 4hour, 6hour, 8hour, 10hour, 12hour
  AUC of Nintedanib and DWN12088

CONTACTS AND LOCATIONS:
Overall Officials: Kim, Principal Investigator — CHA UNITERSITY BUNDANG MEDICAL CENTER
Locations (1):
- Cha Unitersity Bundang Medical Center, Seongnam-si, South Korea